CLINICAL TRIAL: NCT03602417
Title: Comparison of Flare Type Self-expandable Metal Stent With Conventional D-type Self-expandable Metal Stent for Malignant Colorectal Obstruction
Brief Title: Flare Type Self-expandable Metal Stent for Malignant Colorectal Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Associate Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUH13
Record Dates: First submitted 2017-09-19; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; stent
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flare type stent (Experimental): Flare type stent (Taewoong medical) has a wide diameter at proximal end to prevent stent migration.
  Interventions: Device: Flare type stent
- Conventional D-type stent (Active Comparator): Conventional D-type (Taewoong medical) stent has a same diameter at both ends.
  Interventions: Device: Conventional D-type stent

INTERVENTIONS:
Device: Flare type stent — Flare type has a wide diameter at proximal portion to prevent stent migration.
  Arms: Flare type stent
Device: Conventional D-type stent — This stent is an original full covered stent to treat malignant colorectal obstruction.
  Arms: Conventional D-type stent

SUMMARY:
This study compares flare type self-expandable metal stent with conventional D-type self-expandable metal stent for malignant colorectal obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Malignant colorectal obstruction confirmed by radiologic study

Exclusion Criteria:

* Bowel perforation
* Multiple obstruction
* Benign obstruction
* Pregnancy

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | 48 hours
  Colon obstruction is relieved.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No